CLINICAL TRIAL: NCT05648136
Title: Immune Profile Analysis and Biomarker Identification in Women With Repeated Implantation Failure or Unexplained Recurrent Spontaneous Miscarriage
Acronym: ERIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0077
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Repeated Embryo Implantation Failure; Recurrent Miscarriage; Immune System
Keywords: repeated embryo implantation failure; recurrent spontaneous miscarriage; immunological analysis; immune system
MeSH Terms: conditions — Abortion, Habitual | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): * Women aged 18 to 39 years
  * with a history of RIF or unexplained RM
  * with a negative diagnostic work-up (including pelvic ultrasound and hysteroscopy, parental karyotype, thyroid function test, and anti-thyroid and anti-phospholipid antibodies)
  * with a basal FSH level <10IU/l and AMH level >1.5ng/ml
  * with a regular menstrual cycle of 30+/-5 days
  * receiving a new cycle of in vitro fertilization (IVF) +/- intracytoplasmic sperm injection (ICSI) for patients in the RIF group or a first cycle of IVF +/-ICSI for patients in the RM group
  * received written and oral information and signed an informed consent
  Interventions: Biological: blood sample
- control (Active Comparator): * Controls recruited in the Obstetrics and Gynecology Department with at least one live birth after a spontaneous pregnancy (with a time to conception of less than 12 months for each pregnancy) Voluntary oocyte donors recruited within the CECOS de Picardie (having presented at least one live birth with a delay necessary to conceive of less than 12 months)
  * Controls recruited in the Reproductive Medicine and Biology Department having presented at least one live birth (spontaneous with a delay to conceive of less than 12 months for each pregnancy or after one or two MPA procedures) and benefiting from an IVF+/-ICSI procedure for secondary infertility
  * Controls recruited in the department of Medicine and Reproductive Biology with a normal infertility assessment and benefiting from an IVF procedure with ICSI on male indication.
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Blood sampling by venipuncture will be performed :
  * for patients and controls: between the 20th and 24th day of the menstrual cycle (implantation window) preceding the following IVF+/-ICSI cycle
  * for patients receiving an endometrial biopsy: on the same day as the endometrial biopsy
  * for patients and controls receiving follicular stimulation for ovarian puncture: the day of the oocyte puncture
  * for patients and controls undergoing embryo transfer: on the day of embryo implantation

SUMMARY:
Implantation is a determining step in human reproduction which requires the transition from a pro-inflammatory state to an anti-inflammatory state allowing the implantation of a competent embryo within a receptive endometrium, and then the maternal immunotolerance towards the alloantigenic fetus. Repeat implantation failures (RIFs), that refers to the fail to achieve a clinical pregnancy after the transfer of at least 3-4 good quality embryos or two blastocysts, and unexplained recurrent spontaneous miscarriage (RM) (≥2-3) could be related in some patients to immune imbalances characterized by an excessive and prolonged inflammatory response and/or a defect of anti-inflammatory regulation. In this context, several therapies have been evaluated in patients with RIFs or RMs in order to restore the immune balance, with heterogeneous results. No serum biomarker assay has been routinely approved to identify patients with immune imbalances that may explain repeated pregnancy failures and to predict the success of the subsequent IVF/ICSI cycle. The immunological analysis on peripheral blood will be based on the determination of the proportions of immune subpopulations (e.g. CD4+ et CD8+, TH1, TH2, TH17, Treg, ILC 1, ILC2, and ILC3) on the one hand and the circulating level of plasma cytokines on the other hand.

ELIGIBILITY:
Inclusion Criteria:

* For patients :
* Women aged 18 to 39 years
* women with a history of RIF or unexplained RM
* women with a negative diagnostic work-up (including pelvic ultrasound and hysteroscopy, parental karyotype, thyroid function test, and anti-thyroid and anti-phospholipid antibodies)
* women with a basal FSH level <10IU/l and AMH level >1.5ng/ml
* women with a regular menstrual cycle of 30+/-5 days
* women receiving a new cycle of in vitro fertilization (IVF) +/- intracytoplasmic sperm injection (ICSI) for patients in the RIF group or a first cycle of IVF +/-ICSI for patients in the RM group
* women received written and oral information and signed an informed consent

For control groups:

* Controls recruited in the Obstetrics and Gynecology Department with at least one live birth after a spontaneous pregnancy (with a time to conception of less than 12 months for each pregnancy) Voluntary oocyte donors recruited within the CECOS de Picardie (having presented at least one live birth with a delay necessary to conceive of less than 12 months)
* Controls recruited in the Reproductive Medicine and Biology Department having presented at least one live birth (spontaneous with a delay to conceive of less than 12 months for each pregnancy or after one or two MPA procedures) and benefiting from an IVF+/-ICSI procedure for secondary infertility
* Controls recruited in the department of Medicine and Reproductive Biology with a normal infertility assessment and benefiting from an IVF procedure with ICSI on male indication.

Exclusion Criteria:

* Ongoing pelvic and/or systemic infection
* Chronic infectious endometritis
* Active neoplasia
* Autoimmune and autoinflammatory disease
* Celiac disease
* Thrombophilia (including positive anti-phospholipid antibodies)
* Endocrine pathology (including dysthyroidism and diabetes)
* Endometriosis
* Polycystic ovary syndrome and ovulatory disorders
* Premature ovarian failure
* IVF by oocyte donation
* Tubal obstructions or lesions, uterine and cervical anomalies
* Partners with extreme oligoastheno-spermia and/or sperm DNA fragmentation >30
* Sperm donations
* Patients unable to give informed consent

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 150 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Variation of the proportion of CD4+ subpopulations between both patient groups | 18 months
Variation of the proportion of CD8+ subpopulations between both patient groups | 18 months
Variation of the proportion of TH1 subpopulations between both patient groups | 18 months
Variation of the proportion of TH2 subpopulations between both patient groups | 18 months
Variation of the proportion of TH17 subpopulations between both patient groups | 18 months
Variation of the proportion of Treg subpopulations between both patient groups | 18 months
Variation of the proportion of ILC 1 subpopulations between both patient groups | 18 months
Variation of the proportion of ILC 2 subpopulations between both patient groups | 18 months
Variation of the proportion of ILC 3 subpopulations between both patient groups | 18 months
Variation of the proportion of TNFα concentrations between both patient groups | 18 months
Variation of the proportion of IFN gamma concentrations between both patient groups | 18 months
Variation of the proportion of TGF-β concentrations between both patient groups | 18 months
Variation of the proportion of IL-10 concentrations between both patient groups | 18 months
Variation of the proportion of IL-17 concentrations between both patient groups | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No